CLINICAL TRIAL: NCT00673465
Title: A Randomized, Placebo-controlled, Three-Way Crossover Study to Evaluate the Effect of SCH 497079 on Metabolic Parameters and to Determine the Influence of Race/Ethnic Origin on Therapeutic Response
Brief Title: Effect of SCH 497079 on Metabolic Parameters and Influence of Race/Ethnic Origin on Therapeutic Response (Study P05338)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P05338; MK-7079-007 (Other: Merck protocol number)
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment sequence 1: SCH 497079 → Placebo → Metformin (Experimental): Participants received SCH 497079 daily for 4 weeks followed by placebo daily for 4 weeks followed by metformin daily for 4 weeks.
  Interventions: Drug: SCH 497079; Drug: Placebo; Drug: Metformin
- Treatment sequence 2: Placebo → Metformin → SCH 497079 (Experimental): Participants received placebo daily for 4 weeks followed by metformin daily for 4 weeks followed by SCH 497079 daily for 4 weeks.
  Interventions: Drug: SCH 497079; Drug: Placebo; Drug: Metformin
- Treatment sequence 3: Metformin → SCH 497079 → Placebo (Experimental): Participants received metformin daily for 4 weeks followed by SCH 497079 daily for 4 weeks followed by placebo daily for 4 weeks.
  Interventions: Drug: SCH 497079; Drug: Placebo; Drug: Metformin
- Treatment sequence 4: SCH 497079 → Metformin → Placebo (Experimental): Participants received SCH 497079 daily for 4 weeks followed by metformin daily for 4 weeks followed by placebo daily for 4 weeks.
  Interventions: Drug: SCH 497079; Drug: Placebo; Drug: Metformin
- Treatment sequence 5: Placebo → SCH 49709 → Metformin (Experimental): Participants received placebo daily for 4 weeks followed by SCH 497079 daily for 4 weeks followed by metformin daily for 4 weeks.
  Interventions: Drug: SCH 497079; Drug: Placebo; Drug: Metformin
- Treatment sequence 6: Metformin → Placebo → SCH 497079 (Experimental): Participants received metformin daily for 4 weeks followed by placebo daily for 4 weeks followed by SCH 497079 daily for 4 weeks.
  Interventions: Drug: SCH 497079; Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: SCH 497079 — SCH 497079 100 mg capsule, administered orally, once daily for 4 weeks
Drug: Placebo — Placebo capsules matching SCH 497079, administered orally, once daily for 4 weeks
Drug: Metformin — Metformin extended release 750 mg, 2 tablets administered orally, once daily for 4 weeks (1500 mg total daily dose)

SUMMARY:
The purpose of this study is to evaluate the effect of SCH 497079 on metabolic parameters and to determine the influence of race/ethnic origin on therapeutic response.

DETAILED DESCRIPTION:
This study includes two parts, each part includes three consecutive 28-day treatment periods. Part 1 (to be conducted in the United States): each participant will receive the following treatments for 28 days in each of three treatment periods in an order determined by a random code: SCH 497079, or matching placebo, or metformin.

Part 2 (to be conducted in India): this part of the study will be conducted after completion of Part 1 and an analysis indicates a clinically significant decrease in blood glucose in participants with type 2 diabetes mellitus (T2DM) compared to placebo. The same procedures conducted in Part 1 will be conducted in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age to 65 years of age, of either sex, and having a body mass index (BMI) between 27 and 35, inclusive (USA participants)
* Clinical laboratory tests (complete blood count, blood chemistry, and urinalysis) within normal limits (excluding glucose and other changes usually associated with diabetes eg, dyslipidemia)
* Type 2 diabetes mellitus

Exclusion Criteria:

* Female participants who are premenopausal or are not surgically sterilized. Participants who are pregnant, intend to become pregnant (within 3 months of ending the study), or are breast-feeding.
* Participants who have received insulin therapy within 6 months, prior to Day 1/Period 1 or who require thiazide diuretics, beta-blockers and cyclic hormone therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-04-17 (Actual); Primary Completion 2008-12-11 (Actual); Study Completion 2008-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1 was conducted in the United States. If an analysis at the end of Part 1 demonstrated that SCH 497079 exhibited a clinically significant glucose lowering effect, Part 2 was to be conducted in India. Part 2 of the study was not conducted.
Groups:
- Part 1/Treatment Sequence 1: SCH 497079 → Placebo → Metformin; Part 2/Treatment Sequence 1: SCH 497079 → Placebo → Metformin: Participants received SCH 497079 daily for 4 weeks (Period 1) followed by placebo daily for 4 weeks (Period 2) followed by metformin daily for 4 weeks (Period 3).
- Part 1/Treatment Sequence 2: Placebo → Metformin → SCH 497079: Participants received placebo daily for 4 weeks (Period 1) followed by metformin daily for 4 weeks (Period 2)followed by SCH 497079 daily for 4 weeks (Period 3).
- Part 1/Treatment Sequence 3: Metformin → SCH 497079 → Placebo: Participants received metformin daily for 4 weeks (Period 1) followed by SCH 497079 daily for 4 weeks (Period 2)followed by placebo daily for 4 weeks (Period 3).
- Part 1/Treatment Sequence 4: SCH 497079 → Metformin → Placebo; Part 2/Treatment Sequence 4: SCH 497079 → Metformin → Placebo: Participants received SCH 497079 daily for 4 weeks (Period 1) followed by metformin daily for 4 weeks (Period 2) followed by placebo daily for 4 weeks (Period 3).
- Part 1/Treatment Sequence 5: Placebo → SCH 49709 → Metformin; Part 2/Treatment Sequence 5: Placebo → SCH 49709 → Metformin: Participants received placebo daily for 4 weeks (Period 1) followed by SCH 497079 daily for 4 weeks (Period 2) followed by metformin daily for 4 weeks (Period 3).
- Part 1/Treatment Sequence 6: Metformin → Placebo → SCH 497079: Participants received metformin daily for 4 weeks (Period 1) followed by placebo daily for 4 weeks (Period 2) followed by SCH 497079 daily for 4 weeks (Period 3).
- Part 2/Treatment Sequence 2: Placebo → Metformin → SCH 497079: Participants received placebo daily for 4 weeks (Period 1) followed by metformin daily for 4 weeks (Period 2) followed by SCH 497079 daily for 4 weeks (Period 3).
- Part 2/Treatment Sequence 3: Metformin → SCH 497079 → Placebo: Participants received metformin daily for 4 weeks (Period 1) followed by SCH 497079 daily for 4 weeks (Period 2) followed by placebo daily for 4 weeks (Period 3).
- Part 2/Treatment Sequence 6: Metformin → Placebo → SCH 497079: Participants received metformin daily for 4 weeks (Period 1) followed by placebo daily for 4 weeks(Period 2) followed by SCH 497079 daily for 4 weeks (Period 3).
Period: Part 1/Period 1 (United States)
Arm/Group | Part 1/Treatment Sequence 1: SCH 497079 → Placebo → Metformin | Part 1/Treatment Sequence 2: Placebo → Metformin → SCH 497079 | Part 1/Treatment Sequence 3: Metformin → SCH 497079 → Placebo | Part 1/Treatment Sequence 4: SCH 497079 → Metformin → Placebo | Part 1/Treatment Sequence 5: Placebo → SCH 49709 → Metformin | Part 1/Treatment Sequence 6: Metformin → Placebo → SCH 497079 | Part 2/Treatment Sequence 1: SCH 497079 → Placebo → Metformin | Part 2/Treatment Sequence 2: Placebo → Metformin → SCH 497079 | Part 2/Treatment Sequence 3: Metformin → SCH 497079 → Placebo | Part 2/Treatment Sequence 4: SCH 497079 → Metformin → Placebo | Part 2/Treatment Sequence 5: Placebo → SCH 49709 → Metformin | Part 2/Treatment Sequence 6: Metformin → Placebo → SCH 497079
Started | 3 | 3 | 3 | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1/Period 2 (United States)
Arm/Group | Part 1/Treatment Sequence 1: SCH 497079 → Placebo → Metformin | Part 1/Treatment Sequence 2: Placebo → Metformin → SCH 497079 | Part 1/Treatment Sequence 3: Metformin → SCH 497079 → Placebo | Part 1/Treatment Sequence 4: SCH 497079 → Metformin → Placebo | Part 1/Treatment Sequence 5: Placebo → SCH 49709 → Metformin | Part 1/Treatment Sequence 6: Metformin → Placebo → SCH 497079 | Part 2/Treatment Sequence 1: SCH 497079 → Placebo → Metformin | Part 2/Treatment Sequence 2: Placebo → Metformin → SCH 497079 | Part 2/Treatment Sequence 3: Metformin → SCH 497079 → Placebo | Part 2/Treatment Sequence 4: SCH 497079 → Metformin → Placebo | Part 2/Treatment Sequence 5: Placebo → SCH 49709 → Metformin | Part 2/Treatment Sequence 6: Metformin → Placebo → SCH 497079
Started | 3 | 3 | 3 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1/Period 3 (United States)
Arm/Group | Part 1/Treatment Sequence 1: SCH 497079 → Placebo → Metformin | Part 1/Treatment Sequence 2: Placebo → Metformin → SCH 497079 | Part 1/Treatment Sequence 3: Metformin → SCH 497079 → Placebo | Part 1/Treatment Sequence 4: SCH 497079 → Metformin → Placebo | Part 1/Treatment Sequence 5: Placebo → SCH 49709 → Metformin | Part 1/Treatment Sequence 6: Metformin → Placebo → SCH 497079 | Part 2/Treatment Sequence 1: SCH 497079 → Placebo → Metformin | Part 2/Treatment Sequence 2: Placebo → Metformin → SCH 497079 | Part 2/Treatment Sequence 3: Metformin → SCH 497079 → Placebo | Part 2/Treatment Sequence 4: SCH 497079 → Metformin → Placebo | Part 2/Treatment Sequence 5: Placebo → SCH 49709 → Metformin | Part 2/Treatment Sequence 6: Metformin → Placebo → SCH 497079
Started | 3 | 3 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (India)
Arm/Group | Part 1/Treatment Sequence 1: SCH 497079 → Placebo → Metformin | Part 1/Treatment Sequence 2: Placebo → Metformin → SCH 497079 | Part 1/Treatment Sequence 3: Metformin → SCH 497079 → Placebo | Part 1/Treatment Sequence 4: SCH 497079 → Metformin → Placebo | Part 1/Treatment Sequence 5: Placebo → SCH 49709 → Metformin | Part 1/Treatment Sequence 6: Metformin → Placebo → SCH 497079 | Part 2/Treatment Sequence 1: SCH 497079 → Placebo → Metformin | Part 2/Treatment Sequence 2: Placebo → Metformin → SCH 497079 | Part 2/Treatment Sequence 3: Metformin → SCH 497079 → Placebo | Part 2/Treatment Sequence 4: SCH 497079 → Metformin → Placebo | Part 2/Treatment Sequence 5: Placebo → SCH 49709 → Metformin | Part 2/Treatment Sequence 6: Metformin → Placebo → SCH 497079
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated participants.
Groups:
- All Treated Participants: All participants received SCH 497079 for 4 weeks, placebo for 4 weeks, and metformin for 4 weeks during one of three parts of the study.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
24-hour plasma glucose (AUC/duration) [Mean (Standard Deviation); unit: mg/dL] — Mean 24-hour plasma glucose at baseline. Area under the plasma glucose curve (AUC)/duration is presented as mg/dL and was calculated by dividing AUC (mg/dL*hr) by the duration in hours.
  mg/dL | 207 (34)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamic: Change From Baseline in Mean 24-hour Plasma Glucose (AUC/Duration) at Week 4 (Part 1 - United States)
Description: Change from baseline in 24-hour plasma glucose on the last day of treatment. On the day of the glucose collections (and the day prior to), standardized meals breakfast, lunch, dinner, and snack) were provided and consumed over 15 minutes. AUC/duration is presented as mg/dL and was calculated by dividing AUC (mg/dL*hr) by the duration in hours. Model-based least squares mean: ANOVA extracting the effects due to treatment, sequence, period and participant.
Time Frame: Pre-dose (-30 minutes), pre-standard breakfast (0 hour), 0.5, .75, 1, 2, 3, 4, 4.5, 4.75, 5, 6, 7, 8, 9, 9.5, 9.75, 10, 11, 12, 13, 14, 15, 16, and 24 hours after the beginning of the standardized breakfast on Day -1 and Day 28
Population: All participants who completed study treatment with at least SCH 497079 and placebo.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- SCH 497079: Participants received SCH 497079 daily for 4 weeks during one period of the study.
- Placebo: Participants received placebo daily for 4 weeks during one period of the study.
- Metformin: Participants received metformin daily for 4 weeks during one period of the study.
Arm/Group | SCH 497079 | Placebo | Metformin
Number analyzed (Participants) | 14 | 15 | 14
mg/dL | -4.27 (7.35) | 0.13 (7.09) | -53.8 (7.32)
Statistical Analysis 1: Comparison: SCH 497079 vs Placebo; Test type: Superiority or Other; p = 0.5269, ANOVA; ANOVA model extracting the effect due to treatment, period, sequence and participant; Difference in least squares mean = -4.40, 95% CI 2-sided [-18.5 to 9.7]
Statistical Analysis 2: Comparison: Placebo vs Metformin; Test type: Superiority or Other; p < 0.0001, ANOVA; ANOVA model extracting the effect due to treatment, period, sequence and participant; Difference in least squares mean = -53.9, 95% CI 2-sided [-68.1 to -39.8]

2. Primary Outcome: Pharmacodynamic: Change From Baseline in 24-hour Plasma Glucose (AUC/Duration) at Week 4 (Part 2 - India)
Description: Change from baseline in 24-hour plasma glucose on the last day of treatment. On the day of the glucose collections (and the day prior to), standardized meals (breakfast, lunch, dinner, and snack) were provided and consumed over 15 minutes. AUC/duration is presented as mg/dL and was calculated by dividing AUC (mg/dL*hr) by the duration in hours. Model-based least squares mean: ANOVA extracting the effects due to treatment, sequence, period and participant.
Time Frame: Pre-dose (-30 mnutes), pre-standard breakfast (0 hour), 0.5, .75, 1, 2, 3, 4, 4.5, 4.75, 5, 6, 7, 8, 9, 9.5, 9.75, 10, 11, 12, 13, 14, 15, 16, and 24 hours after the beginning of the standardized breakfast on Day -1 and Day 28
Population: No participants were randomized to treatment during Part 2 of the study.
Arm/Group | SCH 497079 | Placebo | Metformin
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event (Part 1 - United States)
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product, biologic (at any dose), or medical device, which does not necessarily have a causal relationship with the treatment. AEs may include the onset of new illness and the exacerbation of pre-existing conditions.
Time Frame: Up to 14 days after last dose of study drug (up to 98 days)
Population: All randomized participants.
Measure: Number; unit: Participants
Arm/Group | SCH 497079 | Placebo | Metformin
Number analyzed (Participants) | 15 | 16 | 15
Participants | 9 | 6 | 4

4. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event (Part 2 - India)
Description: as for outcome 3
Time Frame: Up to 14 days after last dose of study drug (up to 98 days)
Population: No participants were randomized to treatment during Part 2 of the study.
Arm/Group | SCH 497079 | Placebo | Metformin
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Pharmacodynamic: Change From Baseline in 12-hour Postprandial Plasma Glucose (AUC/Duration) at Week 4 (Part 1 - United States)
Description: The postprandial period is defined as the sum of 4 hours after breakfast, 4 hours after lunch and 4 hours after dinner for a total of 12 hours. AUC/duration is presented as mg/dL and was calculated by dividing AUC (mg/dL*hr) by the duration in hours. Model-based least squares mean: ANOVA extracting the effects due to treatment, sequence, period and participant.
Time Frame: as for outcome 1
Population: All participants who completed study treatment with at least SCH 497079 and placebo.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | SCH 497079 | Placebo | Metformin
Number analyzed (Participants) | 14 | 15 | 14
mg/dL | 0.42 (8.67) | 3.22 (8.35) | -60.3 (8.64)
Statistical Analysis 1: Comparison: SCH 497079 vs Placebo; Test type: Superiority or Other; p = 0.7410, ANOVA; ANOVA model extracting the effect due to treatment, period, sequence and participant; Difference in least squares mean = -2.81, 95% CI 2-sided [-20.1 to 14.5]
Statistical Analysis 2: Comparison: Placebo vs Metformin; Test type: Superiority or Other; p < 0.0001, ANOVA; ANOVA model extracting the effect due to treatment, period, sequence and participant; Difference in least squares mean = -63.6, 95% CI 2-sided [-80.9 to -46.2]

6. Secondary Outcome: Pharmacodynamic: Change From Baseline in 12-hour Postprandial Plasma Glucose (AUC/Duration) at Week 4 (Part 2 - India)
Description: as for outcome 5
Time Frame: as for outcome 1
Population: No participants were randomized to treatment during Part 2 of the study.
Arm/Group | SCH 497079 | Placebo | Metformin
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Pharmacodynamic: Change From Baseline in Plasma Glucose During the 12-hour Post Absorptive State (AUC/Duration) at Week 4 (Part 1 - United States)
Description: The post absorptive state is defined as the remaining part of day and night that is not the postprandial period. The postprandial period is defined as the sum of 4 hours after breakfast, 4 hours after lunch and 4 hours after dinner for a total of 12 hours. AUC/duration is presented as mg/dL and was calculated by dividing AUC (mg/dL*hr) by the duration in hours. Model-based least squares mean: ANOVA extracting the effects due to treatment, sequence, period and participant.
Time Frame: Baseline and Week 4
Population: All participants who completed study treatment with at least SCH 497079 and placebo.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | SCH 497079 | Placebo | Metformin
Number analyzed (Participants) | 14 | 15 | 14
mg/dL | -5.37 (3.85) | -1.78 (3.72) | -28.4 (3.84)
Statistical Analysis 1: Comparison: SCH 497079 vs Placebo; Test type: Superiority or Other; p = 0.3146, ANOVA; ANOVA model extracting the effect due to treatment, period, sequence and participant; Difference in least squares mean = -3.59, 95% CI 2-sided [-10.8 to 3.6]
Statistical Analysis 2: Comparison: Placebo vs Metformin; Test type: Superiority or Other; p < 0.0001, ANOVA; ANOVA model extracting the effect due to treatment, period, sequence and participant; Difference in least squares mean = -26.6, 95% CI 2-sided [-33.8 to -19.4]

8. Secondary Outcome: Pharmacodynamic: Change From Baseline in Plasma Glucose During the 12-hour Post Absorptive State (AUC/Duration) at Week 4 (Part 2 - India)
Description: as for outcome 7
Time Frame: Baseline and Week 4
Population: No participants were randomized to treatment during Part 2 of the study.
Arm/Group | SCH 497079 | Placebo | Metformin
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Pharmacokinetic: Mean Plasma Glucose (Over 24 Hours) at Week 4 (Part 1 - United States)
Description: Blood samples for SCH 497079 pharmacokinetics will be collected at pre-dose/0-hour on Day 1 (Period 1 only) and pre-dose Day 14 and pre-dose/0-hour and at 0.5, 1, 2, 6, 12, and 24 hours post study drug administration (not breakfast) on Day 28 of the placebo and SCH 497079 periods only. In addition to these time points, a sample for metformin level will also be collected pre-dose on Day 1, Day 14, and Day 28 of the metformin administration period only.
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 6, 12, and 24 hours after administration of study drug
Population: No efficacy summary or analysis was completed for this outcome measure since the Part 1 objective was not met (i.e., to determine the 24-hour glycemic profile of type 2 diabetes mellitus [T2DM] participants after four weeks of treatment with SCH 497079 vs. placebo).
Arm/Group | SCH 497079 | Placebo | Metformin
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Pharmacokinetic: Mean Plasma Glucose (Over 24 Hours) at Week 4 (Part 2 - India)
Description: as for outcome 9
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 6, 12, and 24 hours after administration of study drug
Population: No participants were randomized to treatment during Part 2 of the study.
Arm/Group | SCH 497079 | Placebo | Metformin
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Pharmacokinetic: Mean Maximum Observed Plasma Concentration (Cmax) (Part 1 - United States)
Description: as for outcome 9
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 6, 12, and 24 hours after administration of study drug
Population: No efficacy summary or analysis was completed for this outcome measure since the Part 1 objective was not met (i.e., to determine the 24-hour glycemic profile of T2DM participants after four weeks of treatment with SCH 497079 vs. placebo).
Arm/Group | SCH 497079 | Placebo | Metformin
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Pharmacokinetic: Mean Plasma Cmax (Part 2 - India)
Description: as for outcome 9
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 6, 12, and 24 hours after administration of study drug
Population: No participants were randomized to treatment during Part 2 of the study.
Arm/Group | SCH 497079 | Placebo | Metformin
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Pharmacokinetic: Mean Time to Maximum Observed Plasma Concentration (Tmax) (Part 1 - United States)
Description: as for outcome 9
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 6, 12, and 24 hours after administration of study drug
Population: as for outcome 11
Arm/Group | SCH 497079 | Placebo | Metformin
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Pharmacokinetic: Mean Plasma Tmax (Part 2 - India)
Description: as for outcome 9
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 6, 12, and 24 hours after administration of study drug
Population: No participants were randomized to treatment during Part 2 of the study.
Arm/Group | SCH 497079 | Placebo | Metformin
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 14 days after last dose of study drug (up to 98 days)
Description: Of the 17 participants who received at least one dose of study medication, 16 participants received at least one dose of placebo, 15 participants received at least one dose of SCH 497079, and 15 participants received at least one dose of metformin.
Groups:
- Placebo: Participants received placebo daily for 4 weeks during one of 3 parts of the study.
- Metformin: Participants received metformin daily for 4 weeks during one of 3 parts of the study.
Arm/Group | Placebo | SCH 497079 | Metformin
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 6/16 | 9/15 | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | SCH 497079 (N=15) | Metformin (N=15)
Eye haemorrage (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Part 2 of the study was not conducted. Part 2 of the study was to be conducted if the analysis of Part 1 indicated a clinically significant decrease in blood glucose in participants type 2 diabetes mellitus compared to placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the study without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.